CLINICAL TRIAL: NCT05384808
Title: Effects of the Inclusion of a Dog in Psychotherapy on Children's Alliance and Treatment Motivation
Brief Title: Canine-assisted Psychotherapy Motivation Alliance
Acronym: CAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Dr. Karin Hediger, Prof. Dr. Karin Hediger, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-00304
Record Dates: First submitted 2022-05-02; First posted 2022-05-20 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Motivation; Alliance, Therapeutic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No dog present (Experimental): Conventional psychotherapy with no dog being present.
  Interventions: Behavioral: Standard Psychotherapy
- Dog present and active part of therapeutic narrative. (Experimental): The dog is actively integrated into the therapeutic narrative.
  Interventions: Behavioral: Canine-assisted psychotherapy with dog actively integrated.
- Dog present but not active part of therapeutic narrative. (Experimental): The dog is present but not actively integrated into the therapeutic narrative.
  Interventions: Behavioral: Canine-assisted psychotherapy with dog passively integrated.

INTERVENTIONS:
Behavioral: Standard Psychotherapy — Participants receive a standard psychotherapy session with no dog being present.
  Arms: No dog present
Behavioral: Canine-assisted psychotherapy with dog actively integrated. — A dog is present and actively integrated into the therapeutic narrative.
  Arms: Dog present and active part of therapeutic narrative.
Behavioral: Canine-assisted psychotherapy with dog passively integrated. — A dog is present but not actively integrated into the therapeutic narrative.
  Arms: Dog present but not active part of therapeutic narrative.

SUMMARY:
The aim of the study is to investigate the needed extent and the way a dog is integrated into psychotherapeutic interventions for them to be motivating and alliance building for children and adolescents with psychiatric disorders aged 9 to 17 years old. Specifically, we want to elaborate if the dog needs to be integrated into the therapy in a form that it is part of the therapeutic context or if the presence of the dog without being part of the therapeutic context per se is beneficial.

ELIGIBILITY:
Inclusion Criteria for children and adolescents: :

* Age between 9 and 17 years
* Children are seeing the therapist for the first time
* Basic knowledge of child and parents in either German or English to be able to fill in questionnaires
* Informed consent given by legal guardian
* Positive or neutral attitude towards dogs

Exclusion Criteria for children and adolescents: :

* acute psychosis; early childhood autism
* diagnosed developmental disorder or intellectual delay; if not diagnosed, exclusion when questionnaires cannot be completed due to development level
* fear of dogs
* allergic reactions to dogs
* reported aggressive behavior towards animals in the past

Inclusion criteria for therapists:

* working with an own therapy dog
* completed therapy training or if not completed far advanced therapy training under supervision
* working with children and adolescents aged 9 to 17 years

Exclusion criteria for therapists:

* not working with an own therapy dog
* no completed or far advanced therapy training
* not working with children and adolescents aged 9 to 17 years

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic alliance of patients | 9 weeks
  Patient's reported therapeutic alliance is measured after the first, the third and the fifth therapy session of a newly began psychotherapy using the german adaptation of the "Therapeutic Alliance Scales for Children" (TASC)". The TASC consists of 12 items, answered with a 4 point likert scale. The questionnaire assesses the therapeutic alliance from the perception of the child. Four weeks after the fifth therapy session children will be asked to fill in the questionnaire again as follow-up measurement.
Motivation of patients | 9 weeks
  Patient's reported motivation is measured after the first, the third and the fifth therapy session of a newly began psychotherapy using the "Situational Motivation Scale for children (SMS-15)". The SMS-15 consists of 15 items answered with a 7 point likert scale. Four weeks after the fifth therapy session, children will be asked to fill in the questionnaire again as follow-up measurement.

SECONDARY OUTCOMES:
Treatment satisfaction of patients | 4 weeks
  Treatment satisfaction of children is measured after the fifth therapy session as well as four weeks after as follow up using the "treatment assessment questionnaire (FBB)". The FBB consists of 20 items answered with a 5 point likert scale.
Number of missed sessions | 5 weeks
  Number of missed sessions and drop-outs will be documented for each child participating in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Arnskotter W, Martin S, Walitza S, Hediger K. Effects of including a dog on treatment motivation and the therapeutic alliance in child and adolescent psychotherapy: study protocol for a randomized controlled trial. Trials. 2024 Jan 5;25(1):26. doi: 10.1186/s13063-023-07854-4. PMID 38183121